CLINICAL TRIAL: NCT00684697
Title: Double Blind Randomized Placebo Controlled Trial of Iron Supplementation in Premature Infants
Brief Title: Iron Status and Myelination in Premature Infants
Acronym: Piron
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Piron Trial
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Neurodevelopmental Outcome
Keywords: premature infants iron neurodevelopment
MeSH Terms: interventions — Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): low iron dose
  Interventions: Dietary Supplement: iron
- 2 (Active Comparator): intermediate iron dose
  Interventions: Dietary Supplement: iron
- 3 (Experimental): High Iron dose
  Interventions: Dietary Supplement: iron

INTERVENTIONS:
Dietary Supplement: iron — High, intermediate and low iron dosage orally for 2 months

SUMMARY:
Premature infants with iron deficiency if supplemented with more elemental iron than the routine 2mg/kg/day will have improved brain development.

ELIGIBILITY:
Inclusion Criteria:

* Babies less than or equal to 33 weeks gestational age

Exclusion Criteria:

* Infants with cranio-facial malformations
* Torch infections
* Infants with hearing disorders
* Infants receiving erythropoietin
* Infants with subnormal vitamin E levels
* Infants with severe anemia
* Infants who are not on full feeds
* Infant with in-utero exposure to cocaine

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
mean interpeak latency Auditory Neural Myelination | 43-45 weeks PMA
  This will be measured using auditory brain stem response.
mean visual neural myelination | 43-45 weeks PMA
  Visual myelination will be evaluated by visual evoked response.

SECONDARY OUTCOMES:
number of participants with executed function | 3-5 years
  Using a standardize test.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv B Amin, MD MS, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States